CLINICAL TRIAL: NCT06912724
Title: A Cross-Sectional Observational Feasibility Pilot Study in Pediatric Neuroimaging: Quantifying White Matter Microstructural Changes in Adolescents With Multidimensional Assessment of Pubertal Stage
Brief Title: Pediatric Neuroimaging
Status: Recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002396; 002396-AG
Record Dates: First submitted 2025-04-04; First posted 2025-04-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12-19

CONDITIONS: Neurogimaging
Keywords: Pediatric Neuroimaging Pubertal Adolescents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Male and female ages 9-14

SUMMARY:
Background:

Puberty is a normal part of life. Many big changes occur in all parts of the body as a child matures into an adult. Researchers in this study want to find out more about how the brain changes during puberty.

Objective:

To study changes that occur in the brain before, during, and after puberty.

Eligibility:

Healthy children aged 9 to 14 years.

Design:

Participants will have 2 clinic visits. Each visit will last up to 4 hours.

In the first visit, participants will be screened:

They will have a physical exam with blood tests.

They will complete a mental health questionnaire on a computer.

They will undergo a mock magnetic resonance imaging (MRI) scan. Participants will be made comfortable as they lie on the table and slide into the big tube. They will learn what it feels and sounds like to lie still inside a real MRI.

At the second visit, participants will have more tests:

They will have a physical exam with blood tests. This time the doctor will check for their stage of puberty. The doctor will look at and touch their genitals and breasts.

They will have a real MRI exam.

An x-ray will be taken of their hand and wrist. This will show how their bones are maturing.

They will have a DEXA scan. They will lie on a table while a machine uses x-rays to measure the makeup of their bodies, including bone, muscle, and fat.

They will have a 3D body scan. They will wear tight clothes and a shower cap. They will stand on a platform while sensors take pictures of their body.

DETAILED DESCRIPTION:
Study Description:

We aim to establish the feasibility of recruitment of children aged 9 to 14 years old to obtain high-quality neuroimaging of white matter determinants employing the Bayesian Monte Carlo analysis of multicomponent driven equilibrium single-component observation of T1 and T2 (BMC-mcDESPOT) and constrained neurite orientation dispersion and density imaging (C-NODDI) Magnetic Resonance Imaging (MRI) techniques with a cross-sectional observational pilot study. We additionally aim to establish the feasibility of multidimensional assessment of pubertal status and body composition as they relate to brain white matter. Data from this pilot study would inform the design of our intended future longitudinal investigations gathering reference data descriptive of normative cerebral microstructural changes in a healthy young population.

Objectives:

The primary objective is to demonstrate feasibility of obtaining highquality BMC-mcDESPOT and C-NODDI MRI data from participants between 9 and 14 years old.

The main exploratory objective is to demonstrate the feasibility of completing multidimensional assessments of pubertal status and body composition of participants between 9 and 14 years old to be related to the neuroimaging.

Additional exploratory objectives include investigation of associations of neuroimaging parameters with proteomic and metabolomic biomarkers. We will explore the feasibility of Magnetic Resonance Spectroscopy in this cohort. Biomarkers would include markers for brain cell integrity (mainly oligodendrocytes, but also neurons and other glia) in the soluble phase of plasma and associated with plasma Extracellular Vesicles (EVs), to determine the value of including such parameters in any future longitudinal study.

Endpoints:

The primary endpoint is to obtain high-quality BMC-mcDESPOT and C-NODDI MRI data from up to 30 female and up to 30 male participants between 9 and 14 years old.

The main exploratory endpoint is to complete multidimensional assessments of pubertal status and body composition of up to 30 male and up to 30 female participants between ages 9 and 14 years old.

Additional exploratory endpoints are high-quality MRS images and acquisition of proteomic and metabolomic biomarkers for brain cell integrity in the soluble phase of plasma and plasma EVs.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, 9 to 14 years of age.
* In good general health
* Ability of parent/guardian to understand and the willingness to sign a written informed consent document.
* Ability of participant to participate in the assent process and willingness to sign a written informed assent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Any known brain abnormalities (e.g. tumor, periventricular leukomalacia, microcephaly) or history of medical conditions known to affect cerebral micro or macro-structural integrity (e.g., epilepsy, history of stroke, head injury with a loss of consciousness of one hour or more).
* History neurodevelopmental delay or disorder, learning disability, intellectual disability (formerly referred to as mental retardation), autism spectrum disorders, and attention deficit/hyperactivity disorder (ADHD)), as evaluated history, physical and by the SDQ, and if indicated, the KSADS
* History of psychiatric disorder as evaluated by history and the SDQ, and if indicated, the KSADS.
* History of prematurity (< 32 weeks gestational age).
* History of endocrine abnormalities, including diagnosed disorders of thyroid, growth, and precocious or delayed puberty
* History of major medical conditions or chronic medical conditions. Examples include neurological disorders, medical or genetic conditions with associated neurological manifestations, malnutrition, conditions raising risk of micronutrient or macronutrient deficiencies (e.g. inflammatory bowel disease), untreated chronic anemia, cardiovascular disease, significant lung disease (e.g. bronchiectasis), significant liver disease, significant kidney disease, significant autoimmune condition, and chronic infections (e.g. HIV, hepatitis B).
* Pregnancy.
* Not eligible to have an MRI as per the MRI eligibility form and the safety standards of the NIA 3T MRI center.
* Presence of hardware (e.g. orthodontic braces) that may interfere with MRI data quality.
* Any other condition which in the investigator s opinion may adversely affect the subject s ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We aim to recruit up to 80 participants between the ages of 9 and 14 years old over a 1-year period with the goal of completion of all study activities by up to 30 male and up to 30 female participants. Recruitment will occur primarily in the Baltimore, Maryland area, as well as the District of Columbia and Virginia areas.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to obtain high-quality BMC-mcDESPOT and C-NODDI MRI data from up to 30 female and up to 30 male participants between 9 and 14 years old. | 1 year of recruitment
  Number of participants with high-quality BMC-mcDESPOT and C-NODDI MRI data

CONTACTS AND LOCATIONS:
Overall Officials: Tina Gupta, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002396-AG.html